CLINICAL TRIAL: NCT01079637
Title: Midfoot Fusion Bolt (MFB). A Randomized Controlled Multicenter Study to Assess the Effectiveness of Surgical Treatment With Midfoot Fusion Bolt in the Early Stage of Diabetic-neuropathic Charcot Feet
Brief Title: Midfoot Fusion Bolt (MFB) in the Early Stage of Diabetic-neuropathic Charcot Feet
Acronym: MFB
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was stopped because there were not enough eligible patients to complete the study.
Sponsor: AO Clinical Investigation and Publishing Documentation (Other)
Responsible Party: Sponsor
Organization: AO Innovation Translation Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MFB 2010
Record Dates: First submitted 2010-03-01; First posted 2010-03-03 (Estimated); Last update posted 2021-07-28 (Actual); Status verified 2015-06

CONDITIONS: Diabetes Mellitus 1 or 2; Midfoot Charcot Neuroarthropathy
Keywords: Sella and Barrete Stage 0 1 or 2
MeSH Terms: interventions — Surgical Procedures, Operative

ARMS (2):
- Midfoot Fusion Bolt (Experimental)
  Interventions: Procedure: Surgery with Midfoot Fusion Bolt
- Cast treatment (Experimental)
  Interventions: Procedure: Cast treatment

INTERVENTIONS:
Procedure: Surgery with Midfoot Fusion Bolt — Surgery with Midfoot Fusion Bolt
  Arms: Midfoot Fusion Bolt
Procedure: Cast treatment — Cast treatment
  Arms: Cast treatment

SUMMARY:
Randomized clinical trial (RCT) to compare treatment failure rates of surgical arthrodesis with MFB against cast treatment in patients suffering from early stage Charcot neuroarthropathy (CN) of the midfoot (Sella and Barrette stages 0, 1 or 2) within the first 2 years after initial treatment. Treatment failure is defined as the occurrence of one or more of the following: 1. Amputation, 2. Occurrence of ulcer or worsening of existing ulcer, 3. Surgical intervention for correction of deformity after initial treatment. The secondary aims are to compare foot function, radiologic outcome, quality of life, complications and foot temperature between the two groups.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Patients with Diabetes Mellitus Type I or II
* CN stages 0, 1 or 2 of the midfoot (Sella and Barrette classification)
* Willingness and ability to participate in the study follow-up according to the protocol
* Ability to understand and read local language at elementary level
* Signed informed consent

Exclusion Criteria:

* Legal incompetence
* Previous Charcot foot on the affected side
* Active osteomyelitis in the affected foot
* Above knee amputation on the contralateral side
* Patient health status not adequate for surgery
* Active malignacy
* Severe peripheral arterial disease (ankle-brachial index <0.7 or absent digital waveforms on Doppler)
* Ulcer grade 2 or more on the Wagner classification system
* Alcohol or drug abuse
* Life-threatening co-morbidities

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2010-05; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
treatment failure rate | baseline, 3 weeks, 6 weeks, 12 weeks, 6 months, 12 months, 24 months
  Treatment failure is defined as the occurrence of one or more of the following:
  1. Amputation
  2. Occurrence of ulcer or worsening of existing ulcer (according to Wagner classification)
  3. Surgical intervention for correction of deformity after initial treatment

SECONDARY OUTCOMES:
Foot function | baseline, 3 weeks, 6 weeks, 12 weeks, 6 months, 12 months, 24 months
  Foot and ankle ability measure score and standard Range of motion measurements.
Radiologic outcome | baseline, 12 weeks, 12 months
  Weightbearing or simulate lateral and AP x-Rays of both feet will be taken. Talus-first metatarsal and Calcaneus-fifth metatarsal angle will be measured.
Evaluation of the generic quality of life including mobility, self-care, usual activities, pain/discomfort, and anxiety/depression | baseline, 3 weeks, 6 weeks, 12 weeks, 6 months, 12 months, 24 months
  EuroQoL5 questionnaire
Rate of complications | baseline, 3 weeks, 6 weeks, 12 weeks, 6 months, 12 months, 24 months
Foot temperature | baseline, 3 weeks, 6 weeks, 12 weeks, 6 months, 12 months, 24 months
  Diabetica Solutions thermometer

CONTACTS AND LOCATIONS:
Locations (1):
- Dept. of Trauma and Reconstructive Surgery, University of Rostock, Rostock, Germany